CLINICAL TRIAL: NCT03300570
Title: Phase I Double-Blind, Placebo-Controlled Trial of 27 mg Dolcanatide (SP-333) to Demonstrate Colorectal Bioactivity in Healthy Volunteers
Brief Title: Dolcanatide in Preventing Colorectal Cancer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2017-01783; NCI-2017-01783 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00042; MAY2017-09-01 (Other: Mayo Clinic in Rochester); MAY2017-09-01 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-03 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dolcanatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (dolcanatide) (Experimental): Participants receive dolcanatide PO QD for 7 days.
  Interventions: Drug: Dolcanatide; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm B (placebo) (Placebo Comparator): Participants receive placebo PO QD for 7 days.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Dolcanatide — Given PO
  Other Names: SP 333; SP-333; SP333
  Arms: Arm A (dolcanatide)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm B (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies how well dolcanatide works in preventing colorectal cancer in healthy participants. Dolcanatide is similar to a natural hormone released into the intestine. It is thought that people who have low levels of the hormone are more likely to get colon cancer. It may be possible to prevent colon cancer by giving a drug that is similar to the hormone, such as dolcanatide.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the ability of dolcanatide (SP333), when administered as a single daily dose of 27 mg x 7 days, to induce a direct pharmacological effect on cGMP levels, based on biopsy samples from the rectum obtained pre- and post-intervention, as compared to placebo.

SECONDARY OBJECTIVES:

I. To assess the pharmacodynamic (PD) response rate between arms (dolcanatide versus placebo).

II. To confirm the safety and tolerability of dolcanatide, as compared to placebo.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants receive dolcanatide orally (PO) once daily (QD) for 7 days.

ARM B: Participants receive placebo PO QD for 7 days.

After completion of study, participants are followed up at 21 and 51 days.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION
* Able to understand and willingness to sign a written informed consent document and follow study procedures
* Willing to abstain from grapefruit juice during study
* Willing to employ adequate contraception for men and women of childbearing potential; Note: acceptable methods include double barrier methods, intrauterine device (IUD), postmenopausal status documented by serum follicle stimulating hormone (FSH), and/or documentation of surgical sterilization
* Willing to provide blood and tissue specimens for research purposes
* REGISTRATION INCLUSION
* Normal organ function and have normal laboratory findings without clinically significant findings
* Leukocytes >= 3 x 10^3/microliter (B/L)
* Absolute neutrophil count >= 1.5 x 10^3/microliter (B/L)
* Platelets >= 100 x 10^3/microliter (B/L)
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal (ULN)
* Creatinine =< institutional upper limit of normal
* Body mass index < 35 kg/m^2
* No findings in the rectum of advanced adenoma, chronic inflammation, or cancer

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION
* Documented history of advanced adenomas (>= 1 cm in maximal diameter, >= 3 in total number, villous morphology, or high-grade dysplasia) or colorectal cancer
* Family history of polyposis syndrome (e.g., familial adenomatous polyposis [FAP], hereditary nonpolyposis colorectal cancer [HNPCC]) or colorectal cancer (first degree relatives younger than 60 years old)
* History of gastroparesis
* History of surgery involving the luminal gastrointestinal (GI) tract, including bariatric surgery; exception: prior appendectomy >= 60 days prior to pre-registration is not an exclusion criterion
* History of celiac disease
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Previous diagnosis of irritable bowel syndrome, chronic constipation, functional bowel disorders, colonic motility disorder, or opioid-induced constipation
* Any malignancy within 3 years of baseline; exception: participants with a history of basal cell or squamous cell skin cancer may be enrolled at the discretion of the investigator
* Currently receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dolcanatide or to any of the excipients
* History of difficulty with sigmoidoscopy or abnormal colorectal anatomy
* Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women
* Current use of laxatives more than 3 times per week
* Current use of >= 5 cigarettes/day
* Current use of >= 3 alcoholic drinks/day
* Use of anti-coagulants or anti-platelet agents within 5 days prior to anticipated sigmoidoscopy; exception: individuals taking aspirin will not be excluded and will not be subject to a wash-out period
* History of bleeding/coagulation problems
* Any medical condition reported by the participant or documented in the medical record that is judged by the investigator to constitute a risk to safe participation
* Known or suspected mechanical gastrointestinal obstruction
* REGISTRATION EXCLUSION
* Sigmoidoscopy finding requiring clinical intervention
* Use of any illicit or illegal substances detected by urinary drug screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Weinberg, Principal Investigator — Mayo Clinic
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 patients were pre-registered, where 10 were screen failures, leaving 27 patients who proceeded to randomization.
Groups:
- Arm A (Placebo): Participants receive placebo PO QD for 7 days. All participants will undergo sigmoidoscopies at baseline and after seven days of daily dosing with placebo.
- Arm B (Dolcanatide): Participants receive dolcanatide PO QD for 7 days. All participants will undergo sigmoidoscopies at baseline and after seven days of daily dosing with dolcanatide.
Period: Overall Study
Arm/Group | Arm A (Placebo) | Arm B (Dolcanatide)
Started (Randomized) | 13 | 14
Completed (Evaluable for the primary endpoint) | 11 | 13
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Inadequate bowel prep | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B (Dolcanatide): Participants receive dolcanatide PO QD for 7 days.All participants will undergo sigmoidoscopies at baseline and after seven days of daily dosing with dolcanatide.
- Total: Total of all reporting groups
Arm/Group | Arm A (Placebo) | Arm B (Dolcanatide) | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.67) | 48.7 (5.72) | 46.6 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 9 | 14 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status = 0 [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Pharmacological Effect on Cyclic Guanosine Monophosphate (cGMP) Levels for Dolcanatide Arm Versus (vs.) Placebo, as Measured by the Differences in Mean cGMP Levels After 7 Days of Intervention
Description: Pharmacological effect on cyclic guanosine monophosphate (cGMP) levels for dolcanatide arm versus (vs.) placebo, where this effect is defined as the arithmetic difference in mean cGMP levels before and after 7 days of dolcanatide from subject biopsies. This represents the increase in cGMP stimulated by 7 days of dolcanatide in an individual subject. The mean cGMP value will be calculated based on 6 biopsies collected from the rectum during a flexible sigmoidoscopy procedure. Each biopsy was analyzed in triplicate using a commercially available EIA kit.
Time Frame: Baseline to 7 days
Population: Only patients who completed the study in the Participant Flow are included in this analysis.
Measure: Mean (Standard Deviation); unit: pmol/mg
Arm/Group | Arm B (Dolcanatide) | Arm A (Placebo)
Number analyzed (Participants) | 13 | 11
pmol/mg | -0.42 (0.43) | -0.22 (0.29)
Statistical Analysis 1: Comparison: Arm B (Dolcanatide) vs Arm A (Placebo); Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pharmacodynamic (PD) Response Rate
Description: Each participant will be assessed for PD response. The calculation is based on the standardized difference in means for the pharmacological effect on cGMP levels at the participant level, where a subject with a z >= 1.645 will be considered a PD responder. A participant with a z < 1.645 will be considered a non-responder. The PD response rate (percentage) of patients are summarized below by arm.
Time Frame: Baseline to 7 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm B (Dolcanatide) | Arm A (Placebo)
Number analyzed (Participants) | 13 | 11
percentage of patients | 0 | 0

3. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Diarrhea Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The overall adverse event rates (percentages) for grade 3 or higher adverse events regardless of attribution to treatment are reported below. The percentages below are summarized for Diarrhea.
Time Frame: Up to 21 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm B (Dolcanatide) | Arm A (Placebo)
Number analyzed (Participants) | 14 | 13
percentage of patients | 7.1 | 0

ADVERSE EVENTS:
Time Frame: Up to 21 days
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Groups:
- Arm A (Placebo): Participants receive placebo PO QD for 7 days. All participants will undergo sigmoidoscopies at baseline and after seven days of daily dosing withplacebo.
Arm/Group | Arm A (Placebo) | Arm B (Dolcanatide)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 4/13 | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Placebo) (N=13) | Arm B (Dolcanatide) (N=14)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 11 (48)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (5)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03300570/Prot_SAP_000.pdf